CLINICAL TRIAL: NCT07405788
Title: A Registration Study on Percutaneous Coronary Intervention for Patients With Myocardial Infarction at Fujian Provincial Hospital
Brief Title: Percutaneous Coronary Intervention for Myocardial Infarction at Fujian Provincial Hospital
Acronym: Fu-AMI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiyang Lin (Other)
Responsible Party: Sponsor-Investigator, Kaiyang Lin, Chief Physician, Fujian Provincial Hospital
Organization: Fujian Provincial Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: k2017-01-012; k2017-01-012 (Other Grant/Funding Number: Ethics Committee of Fujian Provincial Hospital)
Record Dates: First submitted 2025-12-29; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Percutaneous Coronary Intervention (PCI) (Experimental): The main indicators for evaluating the effectiveness and safety of the experimental intervention measures. Participants will receive the new or experimental treatment as stipulated in the trial protocol.
  Intervention measures description: Standard percutaneous coronary intervention (PCI)
  Interventions: Procedure: Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — The culprit vessels for this surgery: LAD, LCX, RCA, LM Number of stents implanted Total number of diseased vessels Postoperative medication use Preoperative TIMI grade of the culprit vessels, postoperative TIMI grade of the culprit vessels TIMI thrombus burden classification High thrombus burden Thrombus size Thrombus aspiration No reflow/slow blood flow Imaging assessment: baseline ejection fraction, left ventricular end-diastolic diameter, left ventricular end-systolic diameter EF values at follow-up, left ventricular end-diastolic diameter, left ventricular end-systolic diameter at follow-up Follow-up dates for cardiac ultrasound Follow-up dates for cardiac magnetic resonance imaging

SUMMARY:
Research Objectives:

This clinical trial aims to evaluate the efficacy and safety of percutaneous coronary intervention (PCI) in patients with myocardial infarction (MI). The primary objective is to determine whether this approach can reduce the incidence of major adverse cardiovascular events (MACE) compared to current conservative treatment.

Research Questions:

This study aims to address the following key questions:

Does standard PCI improve the clinical outcomes of MI patients (such as cardiovascular death, recurrent myocardial infarction, or revascularization due to ischemia-driven vascular reconstruction)? How safe is PCI, especially in terms of bleeding risk, surgical-related complications, or other adverse events? Does PCI have a significant impact on specific secondary endpoints (such as stent thrombosis, hospitalization for heart failure, or quality of life indicators)?

ELIGIBILITY:
1. Inclusion Criteria:

   1. Clinical diagnosis of acute myocardial infarction.
   2. Successful direct or emergency PCI of the infarct-related artery.
   3. Ability to undergo randomization post-PCI.
   4. Ability to understand and voluntarily sign the informed consent form.
2. Exclusion Criteria:

   1. PCI failure (final TIMI flow < grade 2) or presence of untreated severe stenosis.
   2. Planned staged PCI or other cardiac surgery within 3 months.
   3. Cardiogenic shock (Killip class IV), severe structural heart disease, or contraindications to PCI trial intervention.
   4. Active bleeding or high bleeding risk.
   5. Known allergy to the trial drug or its components.
   6. ALT/AST > 3x upper limit of normal (ULN); eGFR < 30 mL/min/1.73 m².
   7. Non-cardiovascular disease with life expectancy < 1 year (e.g., active malignancy).
   8. History of hemorrhagic stroke, or any ischemic stroke/transient ischemic attack within the past 6 months.
   9. Requirement for long-term oral anticoagulation therapy.
   10. Pregnancy, lactation, or women of childbearing potential not using effective contraception.
   11. Current participation in another interventional clinical trial.
   12. Any condition that may affect trial compliance, safety assessment, or result interpretation per investigator judgment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1344 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of participants experiencing related adverse events after percutaneous coronary intervention | From the time of enrollment (baseline) to the 7-year follow-up after the surgery
  Baseline data: Age, gender, height, weight, body mass index, systolic blood pressure at admission, diastolic blood pressure at admission, heart rate, smoking history, past medical history Hospital Admission Situation Perioperative period: The diseased blood vessels, number of stent implants, and biochemical indicators of this surgery; Primary outcome indicators: During hospitalization, the number of related adverse events that occurred in patients around the 7th day after surgery - hematoma at the puncture site, contrast-induced nephropathy, coronary artery dissection, stent thrombosis, etc.
  Hospitalization events: GRACE score, death during hospitalization Continuous follow-up until the last patient was enrolled (from June 2, 2017 to October 23, 2024): All-cause death, MACE1, stroke, recurrent myocardial infarction, stent restenosis, percutaneous coronary intervention, unplanned vascular reconstruction

IPD SHARING:
Plan to Share IPD: Undecided